CLINICAL TRIAL: NCT00005572
Title: Study of Pathogen-Specific Immune Responses and General Immune Competence in Opportunistic Infections
Brief Title: A Comparison of HIV-Infected Patients With and Without Opportunistic (AIDS-Related) Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5067; AACTG A5067
Record Dates: First submitted 2000-04-28; First posted 2001-08-31 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2003-06

CONDITIONS: Cytomegalovirus Infections; Cytomegalovirus Retinitis; Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Lymphocytes; Histoplasmosis; Recurrence; Cytomegalovirus Retinitis; Cell Division; Immunocompetence; Anti-HIV Agents
MeSH Terms: conditions — Cytomegalovirus Infections; Cytomegalovirus Retinitis; Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Histoplasmosis; Recurrence

SUMMARY:
The purpose of this study is to understand how changes in the immune system of HIV-infected patients affect their risk for 3 serious infections: Pneumocystis carinii pneumonia (PCP), cytomegalovirus (CMV) retinitis, or CMV organ disease. The purpose also is to understand how anti-HIV medicines may improve the immune system in these patients. (This purpose reflects a change in the AIDS-related [opportunistic] infections studied.) Presently, HIV-infected patients who have had PCP or CMV disease stay on lifelong therapy to prevent the return of the disease. This study is trying to see if a special lab test can help identify which patients can stop this preventive therapy without having another episode of PCP or CMV organ disease. (This rationale reflects a change in the AIDS-related infections studied.)

DETAILED DESCRIPTION:
To better understand the relationship between immunologic responses, immune reconstitution, and the occurrence of OIs, observational data need to be collected (1) in patients who present with an OI before initiation of potent antiretroviral therapy, (2) in patients with a history of such OIs who have had secondary prophylaxis or maintenance therapy withdrawn and do not develop OI recurrence after potent antiretroviral therapy, and (3) in controls who were exposed to the pathogen of interest but never were at risk for disease because their immunity was not severely compromised. Immunologic comparisons may identify correlates of protection for a group of patients who do not develop an OI after potent antiretroviral therapy-induced immune reconstitution. Conversely, a subpopulation of patients may be identified that lacks critical host factors of protection and is more likely to develop an OI after immune reconstitution, and therefore would benefit from continued prophylaxis, regardless of CD4 cell count.

This study consists of 3 groups and 8 [AS PER AMENDMENT 4/17/01: 6] subgroups. Clinical microbiological data are collected and samples are obtained for immunologic assays (pathogen-specific and general) in all groups at entry (time of OI presentation for Group 1 patients) and at 12 weeks (except Group 3b). Group 1b patients also are evaluated at 24 weeks [AS PER AMENDMENT 4/17/01: The following text has been deleted: and at the time of diagnosis of immune-recovery vitreitis, if it should develop]. [AS PER AMENDMENT 4/17/01: Once patients in Groups 1, 2, and 3a have completed the Week 12 evaluations, they will be off-study.] Blood samples, 1 to 7 days apart, for peripheral blood mononuclear cells (PBMCs), LPA, and inducible cytokine expression of interferon gamma, interleukin-2, interleukin-4, and interleukin-10 are obtained.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible if they:

* Are HIV positive (except Group 3b).
* Are at least 13 years old (consent of parent or guardian required if under 18).
* Patients may be eligible for Group 1a if they:
* Have acute PCP.
* Have never received potent anti-HIV drugs or have not received potent anti-HIV drugs for at least 8 weeks prior to getting PCP.
* Have a CD4 cell count below 200 cells/mm3.
* Patients may be eligible for Group 1b if they:
* Have CMV disease.
* Meet 1 of the following requirements: (1) have never received potent anti-HIV drug containing a protease inhibitor (PI) or a nonnucleoside reverse transcriptase inhibitor (NNRTI), (2) have not received potent anti-HIV drugs for at least 8 weeks before getting CMV disease, or (3) have been on stable anti-HIV therapy for at least 3 months with no new anti-HIV drugs started before CMV disease returned.
* Have a CD4 cell count below 50 cells/mm3 if patient received anti-HIV drugs at any time in the past.
* Have an eye exam (patients with CMV retinitis).
* Patients may be eligible for Group 2a if they:
* Have a history of PCP.
* Are currently receiving potent anti-HIV drugs.
* Have been enrolled in ACTG 888.
* Have been off drugs to prevent PCP for at least 48 weeks prior to study entry.
* Have not developed PCP while on potent anti-HIV drugs.
* Have a CD4 cell count above 200 cells/mm3.
* Patients may be eligible for Group 2b if they:
* Have a history of CMV retinitis.
* Are currently receiving potent anti-HIV drugs.
* Have been off drugs to prevent CMV retinitis for at least 12 weeks prior to study entry.
* Have not developed CMV retinitis while on potent anti-HIV drugs.
* Have a CD4 cell count above 50 cells/mm3.
* Have an eye exam confirming lack of CMV retinitis activity within 28 days before study entry.
* Patients may be eligible for Group 3a if they:
* Are CMV-positive.
* Have never had PCP or CMV disease.
* Have never had a CD4 count below 200 cells/mm3.
* Have never taken medications to prevent PCP or CMV disease.
* Patients may be eligible for Group 3b if they:
* Are HIV-negative.
* Are CMV-positive.
* (The lay eligibility section reflects changes in the AIDS-related infections treated.)

Exclusion Criteria

Patients will not be eligible if they:

* Have received a vaccine within 14 days of study entry or plan to receive one during the study.
* Have taken GM-CSF, any investigational drugs, or any drugs that might affect the immune system within 30 days of study entry or plan to take 1 of these medications during the study. (Prednisone for patients with PCP and G-CSF is allowed.)
* Abuse drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90

CONTACTS AND LOCATIONS:
Overall Officials: Ron D'Amico, Study Chair — Beth Israel Med Ctr
Locations (16):
- United States (16):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Marin County Specialty Clinic, San Rafael, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Children's Mem Hosp Family Cln / Northwestern Univ Med Schl, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington